CLINICAL TRIAL: NCT00768586
Title: Analysis of the Early Development of the Visual Function in Extreme Premature Infants Under 28th Weeks of Gestation. - A Prospective Study to Identify Normal Values of Flash Visual Evoked Potentials in This Population
Brief Title: Analysis of the Early Development of the Visual Function in Extreme Premature Infants Under 28th Weeks of Gestation
Acronym: fVEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Arnold Pollak, MD, PhD, Medical University Vienna, Head of Department of Pediatrics
Other Study IDs: MUVienna
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-09

CONDITIONS: Vision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Extreme premature infants under the 28th week of gestation.

SUMMARY:
The aim of this study is to collect data on the early visual development of extreme premature infants. The method is the measurement of flash visual evoked potentials and the study population includes premature infants under the 28th weeks of gestation, who have normal cranial ultrasound examinations, normal aEEG, no clinical neurological symptoms and who have a normal ophthalmological status.

fVEP measurements were recorded from the first week of life every second week until term.

The fVEP recordings were performed in active sleep, in stable premature infants, who were continuously monitored. The Nihon Kohden Neuropack 8 was used, the stimulus frequency was 0,5 Hz, artefact free averages were analyzed.

The measurements were analyzed according to the presence and absence of known waveforms, their latencies and amplitudes. Longitudinal analysis was performed to analyse the effect of extrauterine visual development on fVEP with growing gestational ages.

ELIGIBILITY:
Inclusion Criteria:

* All premature infants under the 29th week of gestation entering our ward.

Exclusion Criteria:

* Infants with intracranial abnormalities, cerebral malformations, neurological symptoms or known eye pathology.

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants between the 23-29th week of gestation are included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Latency and Amplitude of Visual Evoked Potential waveforms measured in the first week of life than every second week prospectively until term. | Until term

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weninger, MD, PhD., Principal Investigator — MUV
Locations (1):
- Medical University Vienna, Department of Pediatrics, Neonatology, Vienna, Austria